CLINICAL TRIAL: NCT02405091
Title: A Phase 3, Open-Label, Safety and Tolerability Study of NBI-98854 for the Treatment of Tardive Dyskinesia
Brief Title: Safety and Tolerability Study of NBI-98854 for the Treatment of Tardive Dyskinesia
Acronym: Kinect 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-98854-1402
Record Dates: First submitted 2015-03-27; First posted 2015-04-01 (Estimated); Results first posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Tardive Dyskinesia
MeSH Terms: conditions — Tardive Dyskinesia | interventions — valbenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose Group 1 (Experimental): Fixed dose of NBI-98854 administered once daily for 48 weeks
  Interventions: Drug: NBI-98854
- Dose Group 2 (Experimental): Fixed dose of NBI-98854 administered once daily up to 48 weeks
  Interventions: Drug: NBI-98854

INTERVENTIONS:
Drug: NBI-98854

SUMMARY:
Phase 3, open-label, study to evaluate the safety and tolerability of NBI-98854 administered once daily (qd) for a total of 48 weeks of treatment. This study will enroll approximately 150 medically stable male and female subjects with clinical diagnoses of schizophrenia or schizoaffective disorder with neuroleptic-induced TD or mood disorder with neuroleptic-induced TD.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of childbearing potential must agree to use hormonal or two forms of nonhormonal contraception (dual contraception) consistently during the screening, treatment and follow-up periods of the study.
2. Female subjects must not be pregnant.
3. Have one of the following clinical diagnoses for at least 3 months prior to screening: Schizophrenia or Schizoaffective Disorder, or Mood Disorder
4. Have a clinical diagnosis of neuroleptic-induced TD for at least 3 months prior to screening.
5. Have moderate or severe TD
6. If using maintenance medication(s) for schizophrenia or schizoaffective disorder, or mood disorder, be on stable doses.
7. Be in general good health.
8. Have adequate hearing, vision, and language skills to perform the procedures specified in the protocol.
9. Have a negative urine drug screen for amphetamines, barbiturates, benzodiazepine, phencyclidine, cocaine, opiates, or cannabinoids.

Exclusion Criteria

1. Have an active, clinically significant unstable medical condition within 1 month prior to screening.
2. Have a known history of substance dependence, substance (drug) or alcohol abuse.
3. Have a significant risk of suicidal or violent behavior.
4. Have a known history of neuroleptic malignant syndrome.
5. Have a known history of long QT syndrome or cardiac tachy-arrhythmia.
6. Have a cancer diagnosis within 3 years prior to screening (some exceptions allowed).
7. Have received an investigational drug within 30 days before screening or plan to use an investigational drug (other than NBI-98854) during the study.
8. Have a blood loss ≥550 mL or donated blood within 30 days prior to Baseline.
9. Have an allergy, hypersensitivity, or intolerance to tetrabenazine.
10. Are currently pregnant or breastfeeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2015-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (43):
  - Anaheim, California
  - Glendale, California
  - Irvine, California
  - Long Beach, California
  - Los Angeles, California
  - Oakland, California
  - San Bernardino, California
  - San Diego, California
  - Torrance, California
  - Hockessin, Delaware
  - Bradenton, Florida
  - Hialeah, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - North Miami, Florida
  - Orlando, Florida
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Shreveport, Louisiana
  - Natick, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Nashua, New Hampshire
  - Buffalo, New York
  - New York, New York
  - Rochester, New York
  - High Point, North Carolina
  - Dayton, Ohio
  - Oklahoma City, Oklahoma
  - Conshohocken, Pennsylvania
  - Norristown, Pennsylvania
  - Phoenixville, Pennsylvania
  - Scranton, Pennsylvania
  - DeSoto, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Irving, Texas
  - Petersburg, Virginia
  - Seattle, Washington
  - Spokane, Washington
- Canada (4):
  - Vancouver, British Columbia
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- San Juan, Puerto Rico

REFERENCES:
- [Derived] Sajatovic M, Alexopoulos GS, Burke J, Farahmand K, Siegert S. The effects of valbenazine on tardive dyskinesia in older and younger patients. Int J Geriatr Psychiatry. 2020 Jan;35(1):69-79. doi: 10.1002/gps.5218. Epub 2019 Oct 31. PMID 31617235

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants with clinical diagnoses of schizophrenia or schizoaffective disorder or mood disorder with neuroleptic-induced tardive dyskinesia (TD) from 45 centers in North America and Puerto Rico.
Groups:
- Valbenazine 40mg: Participants received valbenazine 40mg capsule once daily for up to 48 weeks.
- Valbenazine 80mg: Participants received valbenazine 40mg once daily for 4 weeks, then 80mg once daily for up to 44 weeks.
- Valbenazine 80/40mg: Participants received valbenazine 40mg once daily for 4 weeks, then 80 mg. Participants who were unable to tolerate the 80 mg dose had a dose decrease to 40 mg capsule once daily for up to 44 weeks.
Period: Overall Study
Arm/Group | Valbenazine 40mg | Valbenazine 80mg | Valbenazine 80/40mg
Started | 49 | 107 | 11
Completed | 20 | 74 | 9
Not Completed | 29 | 33 | 2
Not completed — Adverse Event | 16 | 10 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Noncompliance | 1 | 6 | 2
Not completed — Withdrawal by Subject | 4 | 8 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 5 | 6 | 0
Not completed — Physician Decision | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set: included all participants who are enrolled into the study and received study drug, with the following two exclusions: (a) participants who withdrew from the study and returned all previously dispensed study drug with all doses present, and (b) participants who had no post-baseline data collected
Groups:
- Valbenazine 40mg: Participants received valbenazine 40mg once daily for up to 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Valbenazine 40mg | Valbenazine 80mg | Valbenazine 80/40mg | Total
Number analyzed (Participants) | 45 | 107 | 11 | 163
Age, Continuous [Mean (Full Range); unit: years] | 56.8 [30 to 80] | 57.8 [32 to 82] | 56.3 [42 to 69] | 57.4 [30 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 48 | 5 | 77
  Male | 21 | 59 | 6 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 48 | 1 | 56
  Not Hispanic or Latino | 38 | 59 | 10 | 107
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 0 | 1
  Black or African American | 16 | 31 | 1 | 48
  Caucasian | 26 | 74 | 10 | 110
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Other: Latina | 1 | 0 | 0 | 1
  Other: Mulatto | 0 | 1 | 0 | 1
BMI at Screening [Mean (Full Range); unit: kg/m^2] | 27.80 [18.0 to 40.8] | 28.95 [18.6 to 41.7] | 27.45 [22.2 to 33.3] | 28.53 [18.0 to 41.7]
Primary Psychiatric Diagnosis [Count of Participants; unit: Participants]
  Schizophrenia/schizoaffective | 37 | 76 | 6 | 119
  Mood disorder | 8 | 31 | 5 | 44
Age at Diagnosis [Mean (Full Range); unit: years] — Population: Date of diagnosis was not available for some participants.
  years
    Age at Schizophrenia/Schizoaffective Diagnosis: number analyzed (Participants) | 32 | 69 | 5 | 106
    Age at Schizophrenia/Schizoaffective Diagnosis | 30.9 [14 to 59] | 28.0 [9 to 63] | 26.2 [17 to 45] | 28.8 [9 to 63]
    Age at Mood Disorder Diagnosis: number analyzed (Participants) | 8 | 30 | 4 | 42
    Age at Mood Disorder Diagnosis | 40.6 [32 to 50] | 36.9 [14 to 55] | 28.3 [11 to 62] | 36.8 [11 to 62]
Age at Tardive Dyskinesia Diagnosis [Mean (Full Range); unit: years] — Population: Date of diagnosis was not available for some participants.
  years
    number analyzed (Participants) | 38 | 81 | 10 | 129
    (all) | 47.8 [24 to 73] | 49.2 [16 to 69] | 44.3 [20 to 66] | 48.4 [16 to 73]
Screening BPRS Total Score [Mean (Full Range); unit: score on a scale] — The Brief Psychiatric Rating Scale (BPRS) is a clinician-rated tool designed to assess the severity of psychopathology in participants with schizophrenia and other psychotic disorders (Overall and Gorham, 1962, 1988). The severity of each of the 18 items of the BPRS is rated on a scale of 1 (not present) to 7 (extremely severe) (total score range: 18 to 126). Higher scores represent greater symptom severity.
  score on a scale | 29.2 [19 to 47] | 27.3 [18 to 45] | 28.4 [19 to 45] | 27.9 [18 to 47]
Baseline AIMS Dyskinesia Total Score [Mean (Standard Deviation); unit: score on a scale] — The AIMS Total Dyskinesia Score rates a total of 7 items, rating involuntary movement from 0 (no dyskinesia) to 4 (severe dyskinesia). Items 1 through 7 include facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). The AIMS dyskinesia total score for Items 1-7 ranges from 0 to 28; a higher score reflects increased severity.
  score on a scale | 14.2 (5.5) | 15.0 (4.5) | 12.8 (4.6) | 14.6 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Monitored for Long-Term Safety of Valbenazine
Description: Number of participants monitored for long-term safety through reporting of treatment-emergent adverse events and monitoring of vital signs, clinical laboratory values, and ECG. Summaries of all treatment-emergent AEs, treatment-related AEs, SAEs, and AEs leading to study drug discontinuation were prepared.
Time Frame: 52 weeks
Population: Safety analysis set: includes all participants who were enrolled in the study and received study drug, with the following two exclusions: (a) participants who withdrew from the study and returned all previously dispensed study drug with all doses present, and (b) participants who had no post-baseline data collected
Measure: Count of Participants; unit: Participants
Groups:
- Valbenazine 80/40mg: Participants received valbenazine 40mg once daily for 4 weeks, then 80mg. Participants who were unable to tolerate the 80mg dose had a dose decrease to 40mg capsule once daily for up to 44 weeks.
Arm/Group | Valbenazine 40mg | Valbenazine 80mg | Valbenazine 80/40mg
Number analyzed (Participants) | 45 | 107 | 11
Participants | 45 | 107 | 11

2. Secondary Outcome: Severity of Tardive Dyskinesia (TD) Symptoms Assessed by Abnormal Involuntary Movements Scale (AIMS) Dyskinesia Total Score Change From Baseline at Week 48; On-site AIMS Raters
Description: Severity of TD symptoms assessed by AIMS dyskinesia total score (sum of items 1 through 7), as assessed by On-Site AIMS video raters. The AIMS Total Dyskinesia Score rates a total of 7 items, rating involuntary movement from 0 (no dyskinesia) to 4 (severe dyskinesia). Items 1 through 7 include facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). The AIMS dyskinesia total score for Items 1-7 ranges from 0 to 28; a higher score reflects increased severity.
Time Frame: Baseline and Week 48
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Valbenazine 40mg | Valbenazine 80mg | Valbenazine 80/40mg
Number analyzed (Participants) | 20 | 74 | 9
score on a scale | -10.2 (1.2) | -11.0 (0.5) | -7.2 (2.2)

3. Secondary Outcome: Severity of Tardive Dyskinesia (TD) Symptoms Assessed by Abnormal Involuntary Movements Scale (AIMS) Dyskinesia Total Score Change From Baseline; Central AIMS Video Raters
Description: Severity of TD symptoms assessed by AIMS dyskinesia total score (sum of items 1 through 7), as assessed by the blinded, Central AIMS Video Raters. The AIMS Total Dyskinesia Score rates a total of 7 items, rating involuntary movement from 0 (no dyskinesia) to 4 (severe dyskinesia). Items 1 through 7 include facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). The AIMS dyskinesia total score for Items 1-7 ranges from 0 to 28; a higher score reflects increased severity.
Time Frame: Baseline, Change from Baseline at Week 8, and Change from Baseline at Week 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Valbenazine 40mg | Valbenazine 80mg | Valbenazine 80/40mg
Number analyzed (Participants) | 45 | 107 | 11
score on a scale
  At Baseline | 10.2 (0.6) | 10.0 (0.4) | 9.3 (0.8)
  Change from Baseline at Week 8: number analyzed (Participants) | 33 | 101 | 10
  Change from Baseline at Week 8 | -4.5 (0.7) | -3.5 (0.4) | -4.9 (1.2)
  Change from Baseline at Week 52: number analyzed (Participants) | 20 | 73 | 9
  Change from Baseline at Week 52 | -1.8 (1.0) | -3.3 (0.5) | 0.2 (1.3)

4. Secondary Outcome: Severity of Tardive Dyskinesia (TD) Symptoms Assessed by Abnormal Involuntary Movements Scale (AIMS) Dyskinesia Total Score Change From Baseline; On-Site AIMS Raters
Description: Severity of TD symptoms assessed by AIMS dyskinesia total score (sum of items 1 through 7), as assessed by On-Site AIMS raters. The AIMS Total Dyskinesia Score rates a total of 7 items, rating involuntary movement from 0 (no dyskinesia) to 4 (severe dyskinesia). Items 1 through 7 include facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). The AIMS dyskinesia total score for Items 1-7 ranges from 0 to 28; a higher score reflects increased severity.
Time Frame: Baseline, Change from Baseline at Week 8, and Change from Baseline at Week 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Valbenazine 40mg | Valbenazine 80mg | Valbenazine 80/40mg
Number analyzed (Participants) | 45 | 107 | 11
score on a scale
  At Baseline | 14.2 (0.8) | 15.0 (0.4) | 12.8 (1.4)
  Change from Baseline at Week 8: number analyzed (Participants) | 33 | 105 | 11
  Change from Baseline at Week 8 | -7.1 (1.0) | -5.4 (0.5) | -7.4 (1.6)
  Change from Baseline at Week 52: number analyzed (Participants) | 20 | 74 | 9
  Change from Baseline at Week 52 | -3.8 (1.2) | -4.6 (0.7) | -3.3 (1.8)

5. Secondary Outcome: Clinical Global Impression - Global Improvement of Tardive Dyskinesia (CGI-TD) at Week 48
Description: Clinician's perspective of the participant's overall improvement of TD symptoms since initiation of study drug dosing. The CGI-TD is based on a 7-point scale (range: 1=very much improved to 7=very much worse).
Time Frame: Week 48
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Valbenazine 80mg: Participants received valbenazine 40mg capsule once daily for 4 weeks, then 80mg once daily for up to 44 weeks.
Arm/Group | Valbenazine 40mg | Valbenazine 80mg | Valbenazine 80/40mg
Number analyzed (Participants) | 20 | 74 | 9
score on a scale | 1.7 (0.2) | 1.6 (0.1) | 2.3 (0.4)

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Description: Adverse events were evaluated at regular study visits throughout the study.
  Events with an onset date during the first four weeks of the NBI-98854 treatment period will be summarized separately from events that occur after the Week 4 visit, as all subjects receive the same dose of 40 mg during the first 4 weeks of treatment. Events with an onset date during the NBI-98854 treatment period after Week 4 will be summarized by treatment group.
Groups:
- Valbenazine 40 mg Through Week 4: Participants received valbenazine 40mg capsule once daily for 4 weeks.
- Valbenazine 40mg Week 4 Through Week 52: Participants received valbenazine 40mg capsule once daily for up to 44 weeks from Week 4 through Week 48.
- Valbenazine 80mg Week 4 Through Week 52: Participants received valbenazine 80mg once daily for up to 44 weeks from Week 4 through Week 48.
- Valbenazine 80/40mg Week 4 Through Week 52: Participants who were unable to tolerate the 80mg dose had a dose decrease to 40mg capsule once daily for up to 44 weeks from Week 4 through Week 48.
Arm/Group | Valbenazine 40 mg Through Week 4 | Valbenazine 40mg Week 4 Through Week 52 | Valbenazine 80mg Week 4 Through Week 52 | Valbenazine 80/40mg Week 4 Through Week 52
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/35 | 1/107 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/163 | 3/35 | 17/107 | 1/11
Other Adverse Events (participants affected / at risk) | 0/163 | 5/35 | 15/107 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valbenazine 40 mg Through Week 4 (N=163) | Valbenazine 40mg Week 4 Through Week 52 (N=35) | Valbenazine 80mg Week 4 Through Week 52 (N=107) | Valbenazine 80/40mg Week 4 Through Week 52 (N=11)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 2 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0
Foreign body trauma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 — Dose at time of Joint dislocation event for Valbenazine 80/40mg Week 4 Through Week 52 group was 40 mg.
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hyponatraemic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Sedation (Nervous system disorders) | 0 | 0 | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valbenazine 40 mg Through Week 4 (N=163) | Valbenazine 40mg Week 4 Through Week 52 (N=35) | Valbenazine 80mg Week 4 Through Week 52 (N=107) | Valbenazine 80/40mg Week 4 Through Week 52 (N=11)
Urinary tract infection (Infections and infestations) | 0 | 3 | 9 | 1 — Dose at time of Urinary tract infection event for Valbenazine 80/40mg Week 4 Through Week 52 group was 40 mg.
Headache (Nervous system disorders) | 0 | 2 | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI has the right to publish results provided such publication does not violate confidentiality or IP provisions within the contract with the Sponsor. Prior to submission for publication or presentation of results, the PI must provide the Sponsor time for review. The Sponsor can request the PI to withhold or remove information from all publications. For a multi-center study, any publication of results by the PI shall not be made before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2015-12-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT02405091/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT02405091/SAP_001.pdf